CLINICAL TRIAL: NCT00472615
Title: Menstrual Effects On Mood Symptoms in Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Dorothy Sit, M.D., Assistant Professor of Psychiatry, University of Pittsburgh, School of Medicine, Department of Psychiatry
Other Study IDs: M01RR000056 (NIH); CMRF of the UPMC Health System
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Menstrual Cycle; Depression; Mania or Hypomania; Predictor
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Background and Rationale for Study: Estrogen and progesterone are female hormones that regulate the menstrual cycle and likely serve an important role in the regulation of mood. Premenstrual Syndrome (PMS) which affects 75% of healthy women is a cyclic pattern of mild dysphoria and physical discomfort that begin 1-2weeks pre-menses, and resolve by 2-3 days post-onset of menses. Up to 66% of women with bipolar disorder (BD) describe premenstrual mood changes that range from mild symptoms to severe worsening that require hospitalization. Therefore, the hormonal shifts of the menstrual cycle likely influence bipolar symptoms, but confirmatory research is lacking.

Study questions: The primary aims and hypotheses are to characterize bipolar mood symptoms throughout the menstrual cycle and to determine if women with BD have: 1) a) increased severity and persistence of depression and mania symptoms in the late luteal (premenstrual) vs early follicular phase, b) larger change in mood symptoms from the late luteal (premenstrual) to the early follicular phase, compared to healthy women, 2) more relapses, in the late luteal compared to the early follicular phase. The secondary aims are to determine: 1) frequency and severity of premenstrual dysphoric disorder (PMDD) type symptoms in bipolar women; 2) association between bipolar mood variability and a) menstrual phase, b) ovulatory vs anovulatory cycles, c) antimanic drug treatment.

DETAILED DESCRIPTION:
Study Design: Women with BD (15 depressed, 15 euthymic), and 15 healthy women will enter the study. Over 3-months, subjects undergo monthly visits to assess mood and function, at the follicular and luteal phases. Ovulation is confirmed with: 1) urine dipstick tests to detect ovulation (LH surge) days8-14 from the onset of menses; 2) serum progesterone levels 7-days post-ovulation (LH surge). Subjects record their mood and physical symptoms on the daily self-report LifeChart and the Daily Rating Form.

Study Population: Women with Bipolar I or II Disorder, between ages 18-45. Primary Outcomes Measures: 1) a) mood severity - scores on the Structured Interview Guide for the Hamilton Depression Scale (SIGHADS) for depression, Mania Rating Scale (MRS) for mania/hypomania, and LifeChart mood ratings depression and mania/hypomania, for the late luteal and early follicular phases; b) persistence of symptoms - proportion of days with mild/moderate/severe depression or mania/hypomania. 2) Relapses - # bipolar episodes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-45;
* Bipolar Disorder (BD) I or II (DSM-IV criteria) must agrees to communication between PI and Psychiatrist;
* Healthy Control without Past or Current Major Depression, Psychotic Disorder, premenstrual syndrome or Premenstrual Dysphoric Disorder;
* 25-31day menstrual cycles;
* Minimum 6 menstrual cycles per year

Exclusion Criteria:

* Current DSM-IV Criteria Alcohol or Substance Abuse/Dependence;
* Pregnancy;
* Chronic Anovulation (<4 menstrual cycles/yr);
* Menopause (< 1menses in 1yr);
* Active thyroid disease;
* Hormonal Contraception

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample and outpatient psychiatric offices
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Sit, M.D., Principal Investigator — University of Pittsburgh, School of Medicine, Department of Psychiatry
Locations (2):
- United States (2):
  - Magee Womens Hospital, UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, School of Medicine, Department of Psychiatry, Pittsburgh, Pennsylvania

REFERENCES:
- See also: Western Psychiatric Institute and Clinic - Women's Behavioral HealthCARE Research Studies — http://www.wpic.pitt.edu/research/wbhc/studies.shtml